CLINICAL TRIAL: NCT04171362
Title: The Effect of Connective Tissue Massage in Patients With Migraine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Yildirim Beyazıt University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019-22.
Record Dates: First submitted 2019-11-18; First posted 2019-11-20 (Actual); Last update posted 2020-09-07 (Actual); Status verified 2019-11

CONDITIONS: Migraine With Aura; Migraine; Migraine Without Aura; Connective Tissue Diseases
MeSH Terms: conditions — Migraine with Aura; Migraine Disorders; Migraine without Aura; Connective Tissue Diseases | interventions — Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Migraine group (Experimental): The study included patients diagnosed by migraine according to International Headache Community criteria with18-65 years of age followed by routine controls and who were volunteered
  Interventions: Other: Connective Tissue Massage; Other: Education
- Control group (Active Comparator): The study included patients diagnosed by migraine according to International Headache Community criteria with 8-65 years of age followed by routine controls and were volunteered
  Interventions: Other: Education

INTERVENTIONS:
Other: Connective Tissue Massage — Connective tissue massage (CTM) is a manipulative technique that facilitates the diagnosis and treatment of a wide range of pathologies. Observation and subsequent manipulation of the skin and subcutaneous tissues can have a beneficial effect upon tissues remote from the area of treatment.
  Arms: Migraine group
Other: Education — Education patients were informed about migraine triggers, migraine prevention and coping strategies and exercise options. The exercises were demonstrated by the physiotherapist

SUMMARY:
The aim of this study was to investigate the effectiveness of connective tissue massage in patients with migraine

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Migraine Disease
* Being volunteer

Exclusion Criteria:

* Serious psychiatric problems with mental and / or communication problems Neurological, inflammatory or endocrine disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2019-03-28 (Actual); Primary Completion 2019-12-10 (Actual); Study Completion 2019-12-20 (Actual)

PRIMARY OUTCOMES:
Migraine Disability Assessment Test | change from baseline at 4 weeks
  To assess the level of disability of patients Migraine Disability Assessment Test (MIDAS) was used. It is a widely used and validated test. MIDAS was translated into Turkish and validity and reliability studies were conducted. MIDAS is a test filled in by patients that identifies migraine disability in all areas of activity during last 3 months.It consists of 5 questions.The total MIDAS score is the sum of the days given as response to these five questions (MIDAS 1 to MIDAS 5). The total score ranges from 0 to 90 and is used to categorize patients in disability grades I to IV. A higher score means more severe disability, placing the patient in a higher disability grade

SECONDARY OUTCOMES:
Pittsburgh Sleep Quality Index | change from baseline at 4 weeks
  Pittsburgh Sleep Quality Index to evaluate sleep quality (PSQI) will be used. It is a reliable and valid scale with 19 questions to assess the presence and severity of the disorder. The questionnaire was adapted to Turkish patients by Ağargün et al. The scale can measure subjective sleep quality, sleep latency, sleep time, sleep efficiency, sleep disturbance, sleep medication use and daytime work. The response of each is scored as 0-3. Having a global score of 5 or higher, indicates bad sleep quality.
Hospital Anxiety and Depression Scale ( | change from baseline at 4 weeks
  Hospital Anxiety and Depression Scale (HADS) will be usedl to assess the anxiety and depression. Validity and reliability of HADS in Turkish was established by Aydemir et al. This scale consists of 14 questions. Half of questions (odd numbers) measures anxiety and the other half (even numbers) measures depression. Answers quartet likert format and are scored between 0-3. The lowest score they can get from the sub-scale is 0, the highest score is 21 for each subscale. 10 point is considered as a treshold for depression and or anxiety.
Nothingham Health Profile | Before the treatment and end of 4 weeks
  Nothingham Health Profile was used to measure quality of life. Nottingham Health Profile, emotional, physical and social problems survey. The Turkish validity was made in 1997 by Küçükdeveci et al.There are 6 sub-sections in the survey which consists of 38 questions in total. These sections include pain (8 questions), physical activity (8 questions),fatigue (3 questions), sleep (5 questions), social isolation (5 questions) and emotional reactions (9 questions) the participant is asked to answer these questions in the form of yes or no. Total score for each section scored as 0-100."0 points" indicates the best health status, "100 points indicates the worst health status.
Allodynia Symptom Checklist | change from baseline at 4 weeks
  To evaluate allodynia symptoms associated with headache attacks "Allodynia Symptom Checklist" will be used. 12 different situations are questioned in this list. Each situations are scored as "does not apply to me", "never", "rarely", "less than half", "half or more often". ITotal score ranged between 0-24 points.

CONTACTS AND LOCATIONS:
Locations (1):
- Özge Çoban, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No